CLINICAL TRIAL: NCT00174200
Title: A Randomized, Double-Blind, Crossover Add-On Study To Assess The Differential Sensitivity Of 2 Spatial Working Memory Tests (The Groton Maze Learning Test [GMLT] And The Motor Delayed Response Test [MDR]) In Non-Agitated, Antipsychotic Drug-Naive First-Episode Schizophrenic Or Schizophreniform Patients Treated With Risperidone 2 Mg Daily Or Placebo
Brief Title: Study To Assess Differential Sensitivity Of 2 Spatial Working Memory Tests In Schizophrenics Treated With Risperidone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A9001229
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Schizophrenia; Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone 2 mg

SUMMARY:
To assess the effect of risperidone 2 mg daily (QD) on the differential sensitivity of 2 spatial working memory tests (the GMLT and MDR) in non-agitated, drug-naive patients suffering from first-episode schizophrenia/schizophreniform disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 50 years old, antipsychotic-naive, non-agitated patients diagnosed with first-episode schizophrenia or schizophreniform disorder.

Exclusion Criteria:

* Evidence or history of clinically significant medical or non-medical impairment that, in the opinion of the investigator, would affect the safety of the patient or interfere with the evaluation of the trial results;
* Patients who have a history of substance (which included alcohol) dependence within 12 months or abuse within 3 months of enrollment, or tested positive for an illicit drug on the Screening urine toxicology test
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2004-12; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Day 8 and change from baseline on Day 15 in performance of the GMLT and MDR tasks.

SECONDARY OUTCOMES:
Additional descriptive analyses: Change from baseline in ESRS, PANSS, SOFAS, SRDEQ, and AVM on D8+15; CGI-C on D8+15
-Change from baseline in GMLT, ODR, ESRS, PANSS, SOFAS, SRDEQ, AVM on D43; CGI-C on D43
-ESRS will also be performed on D4+11

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Canada (2):
  - Pfizer Investigational Site, Dartmouth, Nova Scotia
  - Pfizer Investigational Site, Halifax, Nova Scotia
- Pfizer Investigational Site, Moscow, Russia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001229&StudyName=Study%20To%20Assess%20Differential%20Sensitivity%20Of%202%20Spatial%20Working%20Memory%20Tests%20In%20Schizophrenics%20Treated%20With%20Risperidone